CLINICAL TRIAL: NCT03811964
Title: Study of the Photomotor Reflex to Evaluate the Role of the Non-visual Effects of Light in Neurological, Psychiatric and Ophthalmological Pathologies
Brief Title: Photomotor Reflex to Evaluate the Role of the Non-visual Effects of Light in Neurological, Psychiatric and Ophthalmological Pathologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6791
Record Dates: First submitted 2019-01-09; First posted 2019-01-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Sleep Disorders; Neurological Pathologies; Psychiatric Pathologies; Ophthalmological Pathologies
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- primary sleep-wake disorder (Other): Subjects with primary sleep-wake disorder
  Interventions: Other: Specific light exposures
- neurological pathology (Other): subjects presenting a neurological pathology with disorder of the controls of the wake and the sleep
  Interventions: Other: Specific light exposures
- psychiatric pathology (Other): subject presenting a psychiatric pathology with disorder of the controls of the wake and the sleep
  Interventions: Other: Specific light exposures
- ophthalmological pathology (Other): subject presenting an ophthalmological pathology with possible alteration of the photoreception and / or phototransduction
  Interventions: Other: Specific light exposures
- photosensitivity (Other): subjects with photosensitivity with regulation disorder of sleep and wake
  Interventions: Other: Specific light exposures
- group control (Other): healthy subject
  Interventions: Other: Specific light exposures

INTERVENTIONS:
Other: Specific light exposures — Specific light exposures using light in a wide range of intensities or different light/dark regimens

SUMMARY:
The light has visual and non-visual effects on organism and can act on the behavior, the mood, the cognition and the sleep. These effects are mediated by "classical" retina photoreceptors which allow vision (rods, cones) but also melanopsin cells. The non-visual effects of light seems to be altered in many neurological, psychiatric or ophtalmological conditions but their exact role in the pathogenesis remains poorly understand. The purpose of the study is to increase our knowledge of the non-visual effects of light and establish new therapeutic applications

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged 18 years or older
* Subject having signed a free and informed consent
* Subject affiliated to a social protection scheme Arm 1 :Subjects with primary sleep-wake disorder Arm 2 : subjects presenting a neurological pathology with disorder of the controls of the wake and the sleep Arm 3 : subject presenting a psychiatric pathology pathology with disorder of the controls of the wake and the sleep Arm 4 : subject presenting an ophthalmological pathology with possible alteration of the photoreception and / or phototransduction Arm 5 : subjects with photosensitivity with regulation disorder of sleep and wake Arm 6 : healthy subject

Exclusion Criteria:

Age-Related Macular Degeneration (AMD) and all maculopathies (retinopathies pigmentosa, macular involvement of diabetes)

* Cataract with significant vision loss <5/10
* Chorioretinal neovascularization
* Subject in exclusion period determined by previous or current study
* Impossibility to give the subject information enlightened (subject in emergency situation, difficulties of understanding the subject, ...)
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Pregnancy / Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 726 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
PIPR : Post-Illumination Pupil Response | 1 day
  1 measurement per subject is performed after exposure to monochromatic light exposure

CONTACTS AND LOCATIONS:
Overall Officials: Bourgin Patrice, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No